CLINICAL TRIAL: NCT04306900
Title: Phase 1/1b Study to Evaluate the Safety and Activity of TTX-030 (Anti-CD39) in Combination With Pembrolizumab or Budigalimab and/or Chemotherapy in Subjects With Advanced Solid Tumors
Brief Title: TTX-030 in Combination With Immunotherapy and/or Chemotherapy in Subjects With Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trishula Therapeutics, Inc. (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTX-030-002
Record Dates: First submitted 2020-03-04; First posted 2020-03-13 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor, Adult
Keywords: Gastric (gastroesophageal cancer); Advanced Solid Tumor; Colorectal cancer; Cancer; Metastatic Solid Tumor; Combination Therapy; CD39; Adenosine Pathway; Immunotherapy Immuno-oncology; PD-1 Checkpoint Inhibitor; Docetaxel; Budigalimab; ABBV-181; TTX-030; Non-small cell lung cancer; Urothelial cell cancer; Pancreatic cancer; Pembrolizumab; Keytruda; Bladder cancer; Gemcitabine; Nab-paclitaxel
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Urinary Bladder Neoplasms | interventions — budigalimab; Docetaxel; 130-nm albumin-bound paclitaxel; Gemcitabine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Combo 1 (Experimental): TTX-030 plus budigalimab plus mFOLFOX6
  Interventions: Combination Product: TTX-030, budigalimab and mFOLFOX6
- Combo 2 (Experimental): TTX-030 plus budigalimab plus docetaxel
  Interventions: Combination Product: TTX-030, budigalimab and docetaxel
- Combo 3 (Experimental): TTX-030 plus mFOLFOX6
  Interventions: Combination Product: TTX-030 and mFOLFOX6
- Combo 4 (Experimental): TTX-030 plus pembrolizumab
  Interventions: Combination Product: TTX-030 and pembrolizumab
- Combo 5 (Experimental): TTX-030 plus budigalimab (selected tumors evaluated in expansion)
  Interventions: Combination Product: TTX-030 and budigalimab
- Combo 6 (Experimental): TTX-030 plus budigalimab plus nab-paclitaxel + gemcitabine
  Interventions: Combination Product: TTX-030, budigalimab, nab-paclitaxel and gemcitabine
- Combo 7 (Experimental): TTX-030 plus nab-paclitaxel + gemcitabine
  Interventions: Combination Product: TTX-030, nab-paclitaxel and gemcitabine
- Combo 8 (Experimental): Budigalimab plus mFOLFOX6
  Interventions: Combination Product: Budigalimab and mFOLFOX6

INTERVENTIONS:
Combination Product: TTX-030, budigalimab and mFOLFOX6 — Dose and schedule per protocol
  Arms: Combo 1
Combination Product: TTX-030, budigalimab and docetaxel — Dose and schedule per protocol
  Arms: Combo 2
Combination Product: TTX-030 and mFOLFOX6 — Dose and schedule per protocol
  Arms: Combo 3
Combination Product: TTX-030 and budigalimab — Dose and schedule per protocol
  Arms: Combo 5
Combination Product: TTX-030, budigalimab, nab-paclitaxel and gemcitabine — Dose and schedule per protocol
  Arms: Combo 6
Combination Product: TTX-030 and pembrolizumab — Dose and schedule per protocol
  Arms: Combo 4
Combination Product: TTX-030, nab-paclitaxel and gemcitabine — Dose and schedule per protocol
  Arms: Combo 7
Combination Product: Budigalimab and mFOLFOX6 — Dose and schedule per protocol
  Arms: Combo 8

SUMMARY:
This is a phase 1/1b study of TTX-030 in combination therapy, an antibody that inhibits CD39 enzymatic activity, leading to accumulation of pro-inflammatory adenosine triphosphate (ATP) and reduction of immunosuppressive adenosine, which may change the tumor microenvironment and promote anti-tumor immune response.

This trial will study the safety, tolerability, pharmacokinetics, pharmacodynamics and anti-tumor activity of TTX-030 in combination with immunotherapy and/or standard chemotherapies.

ELIGIBILITY:
Abbreviated Inclusion Criteria:

1. Age 18 years or older, is willing and able to provide informed consent
2. Histologically confirmed diagnosis of unresectable or metastatic solid tumor malignancy in selected tumor types
3. Life expectancy > 12 weeks
4. ECOG performance status of 0-1

Abbreviated Exclusion Criteria:

1. History of allergy or hypersensitivity to study treatment components. Patients with a history of severe hypersensitivity reaction to any monoclonal antibody.
2. Use of investigational agent within 28 days prior to the first dose of study treatment and throughout the study
3. Receiving high-dose systemic steroid therapy or any other form of immunosuppressive therapy
4. History of severe autoimmune disease
5. Uncontrolled intercurrent illness or other active malignancy requiring ongoing treatment

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2024-03-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (26):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - City of Hope Medical Center Clinical Trials Office, Duarte, California
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - Chao Family Comprehensive CC, UCI, Orange, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Sylvester Comprehensive Cancer Center, University of Miami Miller School of Medicine, Miami, Florida
  - Ocala Oncology Center PL, Ocala, Florida
  - Orlando Health UF Health Cancer Center, Orlando, Florida
  - IACT Health - John B. Amos Cancer Center, Columbus, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Nebraska Cancer Center Oncology Hematology West P.C., Omaha, Nebraska
  - Montefiore Medical Center, The Bronx, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Toledo, Toledo, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Prisma-Health Cancer Institute, Greenville, South Carolina
  - West Cancer Center and Research Institute, Germantown, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - NEXT Oncology, San Antonio, Texas
  - Hunstman Cancer Intitute, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Froedtert Hospital & Medical College of Wisconsin, Milwaukee, Wisconsin
- South Korea (6):
  - National Cancer Center, Seogu, Busan
  - National Cancer Center, Ilsandong-gu, Goyang-si, Gyeonggi-do
  - Seoul National University, Seongnam-si Bundan-gu, Gyeonggi-do
  - Samsung Medical Center, Gangnam-gu, Seoul
  - Severance Hospital Yonsei University, Seodaemun-gu, Seoul
  - Asan Medical Center, Songpa-gu, Seoul

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - Safety Lead-in (TTX-030 + Budigalimab + mFOLFOX6): Participants in Cohort 1 were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 20 mg/kg Q2W on Days 1 and 15, plus budigalimab at a dose of 500 mg (Q4W) on Day 1 plus mFOLFOX6 over 48 hours (Q2W) on Day 1 and 15 of each 28-day cycle.
- Cohort 3B - Gastric (TTX-030 + Budigalimab + mFOLFOX6): Participants in Cohort 3B were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 20 mg/kg Q2W on Days 1 and 15, plus budigalimab at a dose of 500 mg (Q4W) on Day 1 plus mFOLFOX6 over 48 hours (Q2W) on Day 1 and 15 of each 28-day cycle.
- Cohort 12 - Gastric (Budigalimab + mFOLFOX6): Participants in Cohort 12 were administered IV budigalimab at a dose of 500 mg (Q4W) on Day 1 plus mFOLFOX6 over 48 hours (Q2W) on Day 1 and 15 of each 28-day cycle.
- Cohort 3A - Gastric (TTX-030 + mFOLFOX6): Participants in Cohort 3A were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 20 mg/kg Q2W on Days 1 and 15 plus mFOLFOX6 over 48 hours (Q2W) on Day 1 and 15 of each 28-day cycle.
- Cohort 2 - mCRPC (TTX-030 + Budigalimab + Docetaxel): Participants in Safety Lead-in Cohort 2 were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 30 mg/kg Q3W plus budigalimab 375 mg Q3W plus docetaxel at a dose of 75 mg/m2 Q3W on Day 1 of each 21-day treatment cycle.
- Cohort 9 - Pancreatic (TTX-030 + Budigalimab + Gemcitabine + Nab-Paclitaxel): Participants in Cohort 9 were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 20 mg/kg Q2W on Days 1 and 15 plus budigalimab at a dose of 500 mg (Q4W) on Day 1 plus gemcitabine 1000 mg/m2 + nab-paclitaxel 125 mg/m2 on Days 1, 8, and 15 each 28-day cycle.
- Cohort 11 - Pancreatic (TTX-030 + Gemcitabine + Nab-Paclitaxel): Participants in Cohort 11 were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 20 mg/kg Q2W on Days 1 and 15 plus gemcitabine 1000 mg/m2 + nab-paclitaxel 125 mg/m2 on Days 1, 8, and 15 each 28-day cycle.
- Cohort 4 - CRC (TTX-030 + Budigalimab): Participants in Cohort 4 were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 30 mg/kg Q3W plus budigalimab at a dose of 375 mg Q3W on Day 1 of each 21-day treatment cycle.
- Cohort 6 - HNSCC (TTX-030 + Budigalimab): Participants in Cohort 6 were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 30 mg/kg Q3W plus budigalimab at a dose of 375 mg Q3W on Day 1 of each 21-day treatment cycle.
- Cohort 8 - GEC (TTX-030 + Budigalimab): Participants in Cohort 8 were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 30 mg/kg Q3W plus budigalimab at a dose of 375 mg Q3W on Day 1 of each 21-day treatment cycle.
- Cohort 10 - UCC (TTX-030 + Pembrolizumab): Participants in Cohort 10 were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 30 mg/kg Q3W plus pembrolizumab at a dose of 200 mg Q3W on Day 1 of each 21-day treatment cycle.
Period: Overall Study
Arm/Group | Cohort 1 - Safety Lead-in (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 3B - Gastric (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 12 - Gastric (Budigalimab + mFOLFOX6) | Cohort 3A - Gastric (TTX-030 + mFOLFOX6) | Cohort 2 - mCRPC (TTX-030 + Budigalimab + Docetaxel) | Cohort 9 - Pancreatic (TTX-030 + Budigalimab + Gemcitabine + Nab-Paclitaxel) | Cohort 11 - Pancreatic (TTX-030 + Gemcitabine + Nab-Paclitaxel) | Cohort 4 - CRC (TTX-030 + Budigalimab) | Cohort 6 - HNSCC (TTX-030 + Budigalimab) | Cohort 8 - GEC (TTX-030 + Budigalimab) | Cohort 10 - UCC (TTX-030 + Pembrolizumab)
Started | 8 | 44 | 25 | 6 | 7 | 28 | 17 | 14 | 5 | 23 | 8
Completed | 8 | 44 | 25 | 6 | 7 | 28 | 17 | 14 | 5 | 23 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 12 - Gastric (Budigalimab + mFOLFOX6: Participants in Cohort 12 were administered IV budigalimab at a dose of 500 mg (Q4W) on Day 1 plus mFOLFOX6 over 48 hours (Q2W) on Day 1 and 15 of each 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Safety Lead-in (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 3B - Gastric (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 12 - Gastric (Budigalimab + mFOLFOX6 | Cohort 3A - Gastric (TTX-030 + mFOLFOX6) | Cohort 2 - mCRPC (TTX-030 + Budigalimab + Docetaxel) | Cohort 9 - Pancreatic (TTX-030 + Budigalimab + Gemcitabine + Nab-Paclitaxel) | Cohort 11 - Pancreatic (TTX-030 + Gemcitabine + Nab-Paclitaxel) | Cohort 4 - CRC (TTX-030 + Budigalimab) | Cohort 6 - HNSCC (TTX-030 + Budigalimab) | Cohort 8 - GEC (TTX-030 + Budigalimab) | Cohort 10 - UCC (TTX-030 + Pembrolizumab) | Total
Number analyzed (Participants) | 8 | 44 | 25 | 6 | 7 | 28 | 17 | 14 | 5 | 23 | 8 | 185
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 31 | 14 | 4 | 4 | 12 | 6 | 9 | 3 | 12 | 3 | 102
  >=65 years | 4 | 13 | 11 | 2 | 3 | 16 | 11 | 5 | 2 | 11 | 5 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (9.40) | 59.5 (12.51) | 63.2 (8.70) | 62.5 (6.28) | 65.7 (7.95) | 65.7 (6.83) | 68.2 (9.5) | 61.4 (10.57) | 65.2 (6.57) | 61 (15.54) | 66.4 (7.42) | 63.1 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 18 | 1 | 2 | 0 | 13 | 6 | 5 | 1 | 8 | 1 | 57
  Male | 6 | 26 | 24 | 4 | 7 | 15 | 11 | 9 | 4 | 15 | 7 | 128
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 25 | 22 | 2 | 0 | 9 | 2 | 2 | 1 | 3 | 3 | 69
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 1 | 0 | 9
  White | 7 | 17 | 3 | 3 | 6 | 16 | 12 | 10 | 3 | 17 | 5 | 99
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 0 | 24 | 21 | 2 | 0 | 8 | 2 | 0 | 1 | 0 | 3 | 61
  United States | 8 | 20 | 4 | 4 | 7 | 20 | 15 | 14 | 4 | 23 | 5 | 124

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as the occurrence of any of the following toxicities within the DLT Evaluation Period if judged by the Investigator and Sponsor to be possibly, probably, or definitely related to TTX-030 or budigalimab.
Time Frame: 7 day load + 1 cycle (1 cycle is 28 days)
Population: Only Cohort 1 and Cohort 2 are the safety lead-in cohorts and were evaluated for DLTs.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2 - mCRPC (TTX-030 + Budigalimab + Docetaxel): Participants in Safety Lead-in Cohort 2 were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 30 mg/kg Q3W plus budigalimab 375mg Q3W plus docetaxel at a dose of 75 mg/m2 Q3W on Day 1 of each 21-day treatment cycle.
Arm/Group | Cohort 1 - Safety Lead-in (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 3B - Gastric (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 12 - Gastric (Budigalimab + mFOLFOX6) | Cohort 3A - Gastric (TTX-030 + mFOLFOX6) | Cohort 2 - mCRPC (TTX-030 + Budigalimab + Docetaxel) | Cohort 9 - Pancreatic (TTX-030 + Budigalimab + Gemcitabine + Nab-Paclitaxel) | Cohort 11 - Pancreatic (TTX-030 + Gemcitabine + Nab-Paclitaxel) | Cohort 4 - CRC (TTX-030 + Budigalimab) | Cohort 6 - HNSCC (TTX-030 + Budigalimab) | Cohort 8 - GEC (TTX-030 + Budigalimab) | Cohort 10 - UCC (TTX-030 + Pembrolizumab)
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Participants | 6 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: The Incident of Adverse Events
Description: Number of study subjects experiencing adverse events (AEs) and serious adverse events (SAEs). Safety profile will be assessed through laboratory evaluations, vital signs, and physical examinations.
Time Frame: Through study completion, an average of 1 year
Population: This set included all participants who received at least 1 dose or any partial dose of study treatment. The Safety Analysis Set was used for safety endpoints and study treatment administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Safety Lead-in (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 3B - Gastric (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 12 - Gastric (Budigalimab + mFOLFOX6) | Cohort 3A - Gastric (TTX-030 + mFOLFOX6) | Cohort 2 - mCRPC (TTX-030 + Budigalimab + Docetaxel) | Cohort 9 - Pancreatic (TTX-030 + Budigalimab + Gemcitabine + Nab-Paclitaxel) | Cohort 11 - Pancreatic (TTX-030 + Gemcitabine + Nab-Paclitaxel) | Cohort 4 - CRC (TTX-030 + Budigalimab) | Cohort 6 - HNSCC (TTX-030 + Budigalimab) | Cohort 8 - GEC (TTX-030 + Budigalimab) | Cohort 10 - UCC (TTX-030 + Pembrolizumab)
Number analyzed (Participants) | 8 | 44 | 25 | 6 | 7 | 28 | 17 | 14 | 5 | 23 | 8
Participants | 8 | 44 | 25 | 6 | 7 | 28 | 17 | 14 | 5 | 23 | 8

3. Secondary Outcome: Confirmed Objective Response Rate (ORR)
Description: ORR is defined as the proportion of subjects with CR or PR.
Time Frame: Through study completion, an average of 1 year
Population: The ORR was defined as the proportion of participants who achieved a BOR of either CR or PR as derived based on the lesion measurement provided by the Investigator per RECIST v1.1. Confirmed ORR was defined as 2 disease response assessments showing objective response (CR or PR) at least 4 weeks apart and was presented with corresponding 2-sided 95% confidence intervals (CIs) based on the Clopper-Pearson method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 - Safety Lead-in (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 3B - Gastric (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 12 - Gastric (Budigalimab + mFOLFOX6) | Cohort 3A - Gastric (TTX-030 + mFOLFOX6) | Cohort 2 - mCRPC (TTX-030 + Budigalimab + Docetaxel) | Cohort 9 - Pancreatic (TTX-030 + Budigalimab + Gemcitabine + Nab-Paclitaxel) | Cohort 11 - Pancreatic (TTX-030 + Gemcitabine + Nab-Paclitaxel) | Cohort 4 - CRC (TTX-030 + Budigalimab) | Cohort 6 - HNSCC (TTX-030 + Budigalimab) | Cohort 8 - GEC (TTX-030 + Budigalimab) | Cohort 10 - UCC (TTX-030 + Pembrolizumab)
Number analyzed (Participants) | 7 | 41 | 23 | 4 | 3 | 27 | 17 | 12 | 5 | 22 | 8
percentage of participants | 14.3 [0.4 to 57.9] | 56.1 [39.7 to 71.5] | 69.6 [47.1 to 86.8] | 75.0 [19.4 to 99.4] | 0 [0.0 to 41.0] | 33.3 [16.5 to 54.0] | 23.5 [6.8 to 49.9] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 52.2] | 9.1 [1.1 to 29.2] | 12.5 [0.3 to 52.7]

4. Secondary Outcome: Best Response (BOR)
Description: The BOR was defined as the best response (in the order of CR, PR, stable disease, and PD) by RECIST 1.1 documented from first dose until the end of study, first disease progression, death, or start of new anticancer therapy, whichever was earliest.
Time Frame: Through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Safety Lead-in (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 3B - Gastric (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 12 - Gastric (Budigalimab + mFOLFOX6) | Cohort 3A - Gastric (TTX-030 + mFOLFOX6) | Cohort 2 - mCRPC (TTX-030 + Budigalimab + Docetaxel) | Cohort 9 - Pancreatic (TTX-030 + Budigalimab + Gemcitabine + Nab-Paclitaxel) | Cohort 11 - Pancreatic (TTX-030 + Gemcitabine + Nab-Paclitaxel) | Cohort 4 - CRC (TTX-030 + Budigalimab) | Cohort 6 - HNSCC (TTX-030 + Budigalimab) | Cohort 8 - GEC (TTX-030 + Budigalimab) | Cohort 10 - UCC (TTX-030 + Pembrolizumab)
Number analyzed (Participants) | 7 | 41 | 23 | 4 | 7 | 27 | 17 | 12 | 5 | 22 | 8
Participants
  CR | 0 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  PR | 1 | 18 | 14 | 3 | 0 | 9 | 4 | 0 | 0 | 1 | 0
  Stable Disease | 2 | 14 | 6 | 0 | 7 | 13 | 10 | 3 | 3 | 5 | 2
  PD | 3 | 2 | 1 | 1 | 0 | 3 | 3 | 8 | 1 | 11 | 5
  NE | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 4 | 0

5. Secondary Outcome: Duration of Response (DOR)
Description: DoR will be defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Time Frame: Through study completion, an average of 1 year
Population: Number (%) of subjects with events (PFS)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3B - Gastric (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 12 - Gastric (Budigalimab + mFOLFOX6) | Cohort 3A - Gastric (TTX-030 + mFOLFOX6) | Cohort 9 - Pancreatic (TTX-030 + Budigalimab + Gemcitabine + Nab-Paclitaxel) | Cohort 11 - Pancreatic (TTX-030 + Gemcitabine + Nab-Paclitaxel) | Cohort 8 - GEC (TTX-030 + Budigalimab) | Cohort 10 - UCC (TTX-030 + Pembrolizumab)
Number analyzed (Participants) | 23 | 16 | 3 | 9 | 4 | 2 | 1
Participants | 13 | 4 | 3 | 4 | 4 | 1 | 0

6. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the proportion of subjects with CR, PR, or SD per RECIST 1.1
Time Frame: Through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Safety Lead-in (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 3B - Gastric (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 12 - Gastric (Budigalimab + mFOLFOX6) | Cohort 3A - Gastric (TTX-030 + mFOLFOX6) | Cohort 2 - mCRPC (TTX-030 + Budigalimab + Docetaxel) | Cohort 9 - Pancreatic (TTX-030 + Budigalimab + Gemcitabine + Nab-Paclitaxel) | Cohort 11 - Pancreatic (TTX-030 + Gemcitabine + Nab-Paclitaxel) | Cohort 4 - CRC (TTX-030 + Budigalimab) | Cohort 6 - HNSCC (TTX-030 + Budigalimab) | Cohort 8 - GEC (TTX-030 + Budigalimab) | Cohort 10 - UCC (TTX-030 + Pembrolizumab)
Number analyzed (Participants) | 7 | 41 | 23 | 4 | 7 | 27 | 17 | 12 | 5 | 22 | 8
Participants | 3 | 37 | 22 | 3 | 2 | 22 | 14 | 3 | 1 | 7 | 1

7. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is measured from documentation of progression or death from any cause, whichever occurs first
Time Frame: Through study completion, an average of 1 year
Population: Participants with events (PFS) by Investigator
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Safety Lead-in (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 3B - Gastric (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 12 - Gastric (Budigalimab + mFOLFOX6) | Cohort 3A - Gastric (TTX-030 + mFOLFOX6) | Cohort 2 - mCRPC (TTX-030 + Budigalimab + Docetaxel) | Cohort 9 - Pancreatic (TTX-030 + Budigalimab + Gemcitabine + Nab-Paclitaxel) | Cohort 11 - Pancreatic (TTX-030 + Gemcitabine + Nab-Paclitaxel) | Cohort 4 - CRC (TTX-030 + Budigalimab) | Cohort 6 - HNSCC (TTX-030 + Budigalimab) | Cohort 8 - GEC (TTX-030 + Budigalimab) | Cohort 10 - UCC (TTX-030 + Pembrolizumab)
Number analyzed (Participants) | 7 | 41 | 23 | 4 | 7 | 27 | 17 | 12 | 5 | 22 | 8
Participants
  PD | 5 | 27 | 9 | 4 | 3 | 14 | 15 | 10 | 3 | 17 | 6
  Death | 1 | 2 | 3 | 0 | 0 | 5 | 2 | 1 | 1 | 2 | 0
  Participants censored | 1 | 12 | 11 | 0 | 4 | 8 | 0 | 1 | 1 | 3 | 2

8. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time interval from the first dose of study treatment to death from any cause. Participants who were lost to follow-up or survived until the end of the study were censored at the last date that they were known to be alive. Medians, Q1, and Q3 of OS and the proportion of participants who were alive at 3, 6, 9, and 12 months from Study Day 1 were derived using KM methods.
Time Frame: Through study completion, an average of 1 year
Population: Participants with events (death)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Safety Lead-in (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 3B - Gastric (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 12 - Gastric (Budigalimab + mFOLFOX6) | Cohort 3A - Gastric (TTX-030 + mFOLFOX6) | Cohort 2 - mCRPC (TTX-030 + Budigalimab + Docetaxel) | Cohort 9 - Pancreatic (TTX-030 + Budigalimab + Gemcitabine + Nab-Paclitaxel) | Cohort 11 - Pancreatic (TTX-030 + Gemcitabine + Nab-Paclitaxel) | Cohort 4 - CRC (TTX-030 + Budigalimab) | Cohort 6 - HNSCC (TTX-030 + Budigalimab) | Cohort 8 - GEC (TTX-030 + Budigalimab) | Cohort 10 - UCC (TTX-030 + Pembrolizumab)
Number analyzed (Participants) | 7 | 41 | 23 | 4 | 7 | 27 | 17 | 12 | 5 | 22 | 8
Participants
  AE | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  PD | 1 | 13 | 4 | 1 | 0 | 9 | 8 | 6 | 1 | 8 | 1
  Other | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  Participants censored | 5 | 28 | 16 | 2 | 7 | 16 | 9 | 5 | 3 | 12 | 7

9. Secondary Outcome: Pharmacokinetics (PK)
Description: Serum concentrations of TTX-030 will be tabulated
Time Frame: Cycles 1-4 (each cycle is 21-28 days)
Population: Pharmacokinetic Parameters of Serum TTX-030 by Treatment and Visit at C1D1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ug/mL)
Groups:
- TTX-030 (Load+Q2W) + Budigalimab (Q4W) + mFOLFOX6 (Q2W): Participants were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 20 mg/kg Q2W on Days 1 and 15, plus budigalimab at a dose of 500 mg (Q4W) on Day 1 plus mFOLFOX6 over 48 hours (Q2W) on Day 1 and 15 of each 28-day cycle.
- TTX-030 (Load+Q2W) + mFOLFOX6 (Q2W): Participants were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 20 mg/kg Q2W on Days 1 and 15 plus mFOLFOX6 over 48 hours (Q2W) on Day 1 and 15 of each 28-day cycle.
- TTX-030 (Load+Q3W) + Budigalimab (Q3W) + Docetaxel (Q3W): Participants were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 30 mg/kg Q3W plus docetaxel at a dose of 75 mg/m2 Q3W on Day 1 of each 21-day treatment cycle.
- TTX-030 (Load+Q2W) + Budigalimab (Q4W) + Gemcitabine + Nab-paclitaxel (Days 1, 8, 15): Participants were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 20 mg/kg Q2W on Days 1 and 15 plus budigalimab at a dose of 500 mg (Q4W) on Day 1 plus gemcitabine 1000 mg/m2 + nab-paclitaxel 125 mg/m2 on Days 1, 8, and 15 each 28-day cycle.
- TTX-030 (Load+Q2W) + Gemcitabine + Nab-paclitaxel (Days 1, 8, 15): Participants were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 20 mg/kg Q2W on Days 1 and 15 plus gemcitabine 1000 mg/m2 + nab-paclitaxel 125 mg/m2 on Days 1, 8, and 15 each 28-day cycle.
- TTX-030 (Load+Q3W) + Budigalimab (Q3W): Participants were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 30 mg/kg Q3W plus budigalimab at a dose of 375 mg Q3W on Day 1 of each 21-day treatment cycle.
- TTX-030 (Load+Q3W) + Pembrolizumab (Q3W): Participants were administered IV TTX-030 at a loading dose of 40 mg/kg 7 days before Cycle 1 Day 1 followed by treatment with 30 mg/kg Q3W plus pembrolizumab at a dose of 200 mg Q3W on Day 1 of each 21-day treatment cycle.
Arm/Group | TTX-030 (Load+Q2W) + Budigalimab (Q4W) + mFOLFOX6 (Q2W) | TTX-030 (Load+Q2W) + mFOLFOX6 (Q2W) | TTX-030 (Load+Q3W) + Budigalimab (Q3W) + Docetaxel (Q3W) | TTX-030 (Load+Q2W) + Budigalimab (Q4W) + Gemcitabine + Nab-paclitaxel (Days 1, 8, 15) | TTX-030 (Load+Q2W) + Gemcitabine + Nab-paclitaxel (Days 1, 8, 15) | TTX-030 (Load+Q3W) + Budigalimab (Q3W) | TTX-030 (Load+Q3W) + Pembrolizumab (Q3W)
Number analyzed (Participants) | 49 | 6 | 7 | 28 | 16 | 41 | 7
(ug/mL) | 503 (39.1) | 449 (24.1) | 814 (26.4) | 511 (28.1) | 458 (15.5) | 601 (41.3) | 679 (31.3)

ADVERSE EVENTS:
Time Frame: Up to 30 days from the last dose of TTX-030, a maximum duration of 2 years of treatment
Description: Safety population = all participants who received at least one dose or any partial dose of TTX-030.
Arm/Group | Cohort 1 - Safety Lead-in (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 3B - Gastric (TTX-030 + Budigalimab + mFOLFOX6) | Cohort 12 - Gastric (Budigalimab + mFOLFOX6) | Cohort 3A - Gastric (TTX-030 + mFOLFOX6) | Cohort 2 - mCRPC (TTX-030 + Budigalimab + Docetaxel) | Cohort 9 - Pancreatic (TTX-030 + Budigalimab + Gemcitabine + Nab-Paclitaxel) | Cohort 11 - Pancreatic (TTX-030 + Gemcitabine + Nab-Paclitaxel) | Cohort 4 - CRC (TTX-030 + Budigalimab) | Cohort 6 - HNSCC (TTX-030 + Budigalimab) | Cohort 8 - GEC (TTX-030 + Budigalimab) | Cohort 10 - UCC (TTX-030 + Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 2/8 | 13/44 | 7/25 | 2/6 | 0/7 | 11/28 | 8/17 | 7/14 | 2/5 | 10/23 | 2/8
Serious Adverse Events (participants affected / at risk) | 4/8 | 27/44 | 16/25 | 2/6 | 4/7 | 16/28 | 8/17 | 4/14 | 2/5 | 10/23 | 3/8
Other Adverse Events (participants affected / at risk) | 8/8 | 43/44 | 25/25 | 6/6 | 7/7 | 28/28 | 17/17 | 14/14 | 1/5 | 23/23 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Safety Lead-in (TTX-030 + Budigalimab + mFOLFOX6) (N=8) | Cohort 3B - Gastric (TTX-030 + Budigalimab + mFOLFOX6) (N=44) | Cohort 12 - Gastric (Budigalimab + mFOLFOX6) (N=25) | Cohort 3A - Gastric (TTX-030 + mFOLFOX6) (N=6) | Cohort 2 - mCRPC (TTX-030 + Budigalimab + Docetaxel) (N=7) | Cohort 9 - Pancreatic (TTX-030 + Budigalimab + Gemcitabine + Nab-Paclitaxel) (N=28) | Cohort 11 - Pancreatic (TTX-030 + Gemcitabine + Nab-Paclitaxel) (N=17) | Cohort 4 - CRC (TTX-030 + Budigalimab) (N=14) | Cohort 6 - HNSCC (TTX-030 + Budigalimab) (N=5) | Cohort 8 - GEC (TTX-030 + Budigalimab) (N=23) | Cohort 10 - UCC (TTX-030 + Pembrolizumab) (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood loss anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic pseudocyst haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic ischaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 10 (10) | 7 (7) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Anuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Safety Lead-in (TTX-030 + Budigalimab + mFOLFOX6) (N=8) | Cohort 3B - Gastric (TTX-030 + Budigalimab + mFOLFOX6) (N=44) | Cohort 12 - Gastric (Budigalimab + mFOLFOX6) (N=25) | Cohort 3A - Gastric (TTX-030 + mFOLFOX6) (N=6) | Cohort 2 - mCRPC (TTX-030 + Budigalimab + Docetaxel) (N=7) | Cohort 9 - Pancreatic (TTX-030 + Budigalimab + Gemcitabine + Nab-Paclitaxel) (N=28) | Cohort 11 - Pancreatic (TTX-030 + Gemcitabine + Nab-Paclitaxel) (N=17) | Cohort 4 - CRC (TTX-030 + Budigalimab) (N=14) | Cohort 6 - HNSCC (TTX-030 + Budigalimab) (N=5) | Cohort 8 - GEC (TTX-030 + Budigalimab) (N=23) | Cohort 10 - UCC (TTX-030 + Pembrolizumab) (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 11 (11) | 1 (1) | 2 (2) | 0 (0) | 5 (5) | 3 (3) | 3 (3) | 0 (0) | 7 (7) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 9 (9) | 5 (5) | 0 (0) | 0 (0) | 7 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 1 (1) | 2 (2) | 5 (5) | 12 (12) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 9 (9) | 7 (7) | 2 (2) | 2 (2) | 15 (15) | 7 (7) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 8 (8) | 5 (5) | 0 (0) | 0 (0) | 9 (9) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 18 (18) | 5 (5) | 3 (3) | 1 (1) | 6 (6) | 6 (6) | 2 (2) | 0 (0) | 7 (7) | 1 (1)
Cough (General disorders) | 0 (0) | 7 (7) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 6 (6) | 1 (1)
COVID-19 (General disorders) | 1 (1) | 10 (10) | 7 (7) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 19 (19) | 8 (8) | 3 (3) | 0 (0) | 10 (10) | 7 (7) | 0 (0) | 0 (0) | 10 (10) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 19 (19) | 6 (6) | 2 (2) | 2 (2) | 10 (10) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema peripheral (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 8 (8) | 4 (4) | 0 (0) | 0 (0) | 6 (6) | 2 (2)
Fatigue (General disorders) | 2 (2) | 17 (17) | 6 (6) | 2 (2) | 7 (7) | 18 (18) | 11 (11) | 2 (2) | 0 (0) | 11 (11) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 28 (28) | 15 (15) | 4 (4) | 3 (3) | 16 (16) | 9 (9) | 3 (3) | 0 (0) | 7 (7) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 16 (16) | 6 (6) | 2 (2) | 2 (2) | 9 (9) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 27 (27) | 17 (17) | 1 (1) | 4 (4) | 12 (12) | 10 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 13 (13) | 8 (8) | 1 (1) | 3 (3) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 4 (4) | 8 (8) | 3 (3) | 1 (1) | 0 (0) | 8 (8) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 11 (11) | 5 (5) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 13 (13) | 3 (3) | 0 (0) | 0 (0) | 10 (10) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT04306900/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT04306900/SAP_001.pdf